CLINICAL TRIAL: NCT05443100
Title: A Non-randomized Pilot Study of the Impact on Rehabilitation Outcomes of a Course of Whole-body Cryostimulation (WBC) Treatment on Patients With Metabolic or Neurological Diseases or Fibromyalgia
Brief Title: Impact of WBC on Patients With Metabolic or Neurological Diseases or Fibromyalgia (WBC-MeNeFi)
Acronym: WBC-MeNeFi
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Auxologico Italiano (Other)
Collaborators: Politecnico di Milano (Other); Università degli Studi di Brescia (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: 31C122
Record Dates: First submitted 2022-06-21; First posted 2022-07-05 (Actual); Last update posted 2025-08-04 (Actual); Status verified 2025-08

CONDITIONS: Obesity; Fibromyalgia; Neurological Conditions
Keywords: Whole-Body cryostimulation; Obesity; Rehabilitation; Catecholamines; Thermal stress
MeSH Terms: conditions — Obesity; Fibromyalgia | interventions — Rehabilitation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rehabilitation (Experimental): Multidisciplinary rehabilitation program consisting of diet and physical exercise for 4 weeks.
  Interventions: Other: Rehabilitation program
- Whole-Body Cryotherapy (Experimental): Rehabilitation program consisting of 10 WBC sessions over two weeks.
  Interventions: Other: Whole-body cryostimulation (WBC); Other: Rehabilitation program

INTERVENTIONS:
Other: Whole-body cryostimulation (WBC) — Multidisciplinary rehabilitation program consisting of 10 WBC sessions.
  Other Names: Whole-body cryotherapy
  Arms: Whole-Body Cryotherapy
Other: Rehabilitation program — Multidisciplinary rehabilitation program consisting of diet and physical exercise.
  Other Names: Multidisciplinary Rehabilitation program

SUMMARY:
The purpose of this clinical trial is to investigate on different types of patients the effects of 10 sessions of whole-body cryostimulation (WBC): 1) in patients with obesity (BMI > 30), we want to investigate whether WBC increases thermogenesis, basal metabolic rate (BMR), respiratory quotient (which indirectly provides an estimate of energy substrate oxidation), reduces chronic inflammatory status, fatigue and pain, and improves functional abilities and general physical and psychological capacities; 2) in patients diagnosed with fibromyalgia and/or osteoarthrytis, we want to investigate the reduction of pain, inflammatory status, increase in functional capacity and general physical and psychological abilities, and improvement in mood; 3) in neurological patients diagnosed with Parkinson's disease, Multiple Sclerosis, and Disimmune Polyneuropathies, the effects of WBC on pain, fatigue, and sleep quality are to be investigated; 4) in normal/overweight (BMI<30 kg/m2) subjects, the effects of WBC on all parameters described previously for the other protocols are to be investigated. Specifically, for all enrolled subjects, we want to assess blood catecholamine levels, investigate the effects of sympathetic response on body composition, blood pressure, heart rate, lipid profile, and physical performance. Three hundred patients admitted for a rehabilitation program (diet + physiotherapy + exercise) will be non-randomly assigned to either a group following the program (R) or a group additionally receiving ten 2-3 minute WBC sessions at -110°C over two weeks (RWBC).

DETAILED DESCRIPTION:
Introduction: Istituto Auxologico Italiano (IAI) has as its institutional mission the study, treatment and rehabilitation of patients with obesity and neurological disorders as well as translational research from bench to bedside to improve these care pathways. The validation of innovative therapeutic modalities of proven efficacy on these patients, potentially scalable to the health care system, is a signature activity of the Institute's Current Research program. IAI in Piancavallo admits 3300 rehabilitation patients with comorbid obesity, including fibromyalgia, and 480 with neurological conditions each year. Pain, chronic fatigue, poor sleep quality, inflammatory status, thymic tone deflection, and obesity have a negative impact on rehabilitation treatment. Whole-body Cryostimulation (WBC) represents an innovative method that induces increased thermogenesis by promoting weight loss, reduced inflammation and oxidative stress with therapeutic effect on fatigue, pain, thymic tone and sleep (Polish Cryomedical Society, Polish Society for Rheumatology). Exposure to cryogenic temperatures would cause activation of the sympathetic system and thus an increase in catecholamine levels, which would stimulate excess adipose tissue to convert from white, metabolically inert tissue to brown, i.e., metabolically active adipose tissue. In fact, it has been previously reported that repeated exposure to WBC reduces inflammation and oxidation, improving immunity, antioxidant activity, and insulin sensitivity, and increasing the percentage of brown adipose tissue (BAT) volume and fatty acid utilization by decreasing the percentage of adipose tissue. This would be reflected in increased tolerance to rehabilitation treatment, improved neuro-cognitive performance and psychological state. The metabolic effect of repeated cold exposure with WBC (browning of adipose tissue and increased thermogenesis) would allow, within multidisciplinary rehabilitation pathways, a better weight loss goal for functional recovery and disease progression in patients with obesity. Since the changes demonstrated at the molecular level after WBC are similar to those induced by exercise, WBC treatment would represent a potential alternative to exercise that is often poorly tolerated in patients with complicated metabolic diseases and disabling neurological conditions and thus a complementary innovative nonpharmacological rehabilitation strategy within a rehabilitation pathway.

Participants: Using a consecutive sampling technique, the investigators will recruit patients for a comprehensive, multidisciplinary rehabilitation program for obesity. Patients of both sex, age 18-65 years with BMI > 35 kg/m2 will be selected and consecutively evaluated for inclusion in the protocol. Exclusion criteria are: severe psychiatric conditions, acute respiratory disease, acute cardiovascular disease, unstable hypertension, cold intolerance, claustrophobia, pregnancy, recent modification of usual drug treatment, previous treatment with WBC, weight loss in the last 3 months, and body temperature greater than 37.5°C. All patients will perform a multidisciplinary rehabilitation program (diet + exercise and physiotherapy).

Study design: Patients will be assigned to either a "rehabilitation + WBC" (RWBC) or "rehabilitation" intervention (R) group in a consecutive, non-randomized manner until the total sample for each group is reached (15 subjects per group).

Anthropometric values, body composition, plasma catecholamine concentration, demographic and hematological analyses, muscle strength and functional values of both groups will be assessed at admission (PRE-T0) and at discharge (POST-T10), two weeks later, for both groups within the hospital facility. They will undergo 10 sessions of WBC over two weeks (1 treatment per day, Monday through Friday, before exercise classes and physical therapy). Skin temperatures will be recorded immediately before and after each WBC exposure. Description of the WBC session: Study participants will be exposed to extremely cold, dry air at -110°C for 2-3 minutes in a cryochamber (Artic, CryoScience, Rome. The first WBC session will last 1 minute at -110°C to familiarize the patient with the cryochamber temperature, while all subsequent treatments will last 2 minutes. The patient's skin surface temperature at the neck, quadriceps, popliteal fossa, and calf will be measured before and after each treatment. The operator supervising the procedure will be in constant visual and vocal contact with the subjects. For safety reasons, the systolic and diastolic blood pressure of each participant will be measured before and after treatment.

Rehabilitation program: The multidisciplinary rehabilitation program will consist of individual nutritional intervention, psychological support, and supervised physical activity throughout hospitalization. All patients will receive a balanced hypocaloric Mediterranean diet with 18-20 % proteins, 27-30 % fats (of which < 8% saturated fat) and 50-55 % carbohydrates (< 15% simple sugars), and 30 g of fibers from fresh vegetables. The diet plan will be organized by the hospital dietitian into three meals: breakfast, lunch, and dinner, with an energy distribution of 20 %, 40 % and 40 %, respectively. Two daily 60-minute physiotherapy sessions consisting of personalized progressive aerobic training, postural control exercises and progressive strengthening exercises were performed under the supervision of a physiotherapist. The first aerobic session performed in the morning after WBC consists of walking at a self-selected cadence. The second session performed in the afternoon consists of arm-cranking at an intensity of 65% of HRmax according to the Karvonen equation ((220 - age) × 0.65).

Measurements. Demographic and clinical characteristics: Baseline demographic and clinical characteristics will be collected at the time of admission and will include age, sex, weight, height and body mass index (BMI).

Body Composition: Body composition will be assessed in the morning in a quiet room at a temperature of 22-25 °C using bioimpedentiometry (BIA) analyzes with the patient in a supine position with lower limbs slightly apart and empty bladder. Whole-body resistance (Rz) and reactance (Xc) will be measured by trained operators and these parameters will be assessed (in Kg and %): fat mass (FM), free fat mass (FFM), muscle mass (MM), appendicular skeletal muscle mass (ASMM).

Skin temperatures: The patient's skin surface temperature (°C) in at the neck,quadriceps, popliteal fossa, and calf will be measured before and after each WBC treatment.

Blood collection and Hematological/Biochemical analyses: Blood samples will be taken in the morning after overnight fasting conditions to determine plasma catecholamine levels (epinephrine, norepinephrine, dopamine, cortisol); red blood cell count (RBC), white blood cell count (WBC), platelet count (PLT), hemoglobin (HGB), hematocrit (HCT), mean corpuscular volume (MCV), mean corpuscular hemoglobin (MCH), mean corpuscular hemoglobin concentration (MCHC), red cell distribution width (RDW), and mean platelet volume (MPV), complete blood count derived inflammatory biomarkers (NLR, dNLR, SII, AISI), erythrocyte sedimentation rate (ESR), C-reactive protein (CRP), TNF-α, cholesterol, HDL, LDL, glucose, insulin.

Performance-based physical functioning: to measure aerobic endurance, we will use the six-minute walk test (6MWT), performed indoors, along a 30-m, flat, undisturbed hospital corridor, with the length scored every 5 m. Chest pain, severe dyspnea, physical exhaustion, muscle cramps, sudden gait instability or other signs of severe distress are additional criteria for stopping the test. The Timed Up and Go test (TUG) test will be used to assess balance and functional mobility. The participant is asked to stand up from a standard chair, walk for 3 minutes, turn around, return to the chair, and sit down. The score corresponds to the time (seconds) taken to perform the test. Isometric strength will be assessed with the hand grip test using the American Society of Hand Therapists (ASHT) protocol as a reference.

Condition specific questionnaires will be administered to assess:

General health: Short-form health survey-36 (SF-36) and World Health Organization Well-being index (WHO5); pain: visual analogue scale (VAS), pain numeric rating scale (PNRS), brief pain inventory (BPI), central sensitization index (CSI), Promis global health scale, the Quantitative Analgesic Questionnaire (QAQ); fatigue: fatigue severity scale (FSS); sleep: Pittsburgh sleep quality index (PSQI), Promis sleep disturbance short form, Epworth Sleepiness Scale; Fibromyalgia Impact Questionnaire (FIQ) for the evaluation of fibromyalgia; Western Ontario and McMaster Universities Osteoarthritis index (WOMAC) for the evaluation for patients with osteoarthritis; psychological weel-being, mood and depression: Psychological General Well-Being Index (PGWBI); State-Trait Anxiety Inventory (STAI); Depression, Anxiety and Stress Scale - 21 Items (DASS-21); Beck's Depression Inventory (BDI); Fear of movement: Tampa Scale of Kinesiophobia (TSK-I); Intestinal function: Wexner score; obesity-related disability: Test of Obesity-Related Disability (SIO Obesity-Related Disability Test, TSD-OC).

Statistical analysis: A sample of 15 obese adult individuals (BMI>35 Kg/m2, age 18-65 years, both sexes) will be considered for each of the two groups, for a total of 30 individuals. Since there is no a priori data on this and it is a pilot study, the sample size was chosen based on the literature, which suggests considering a minimum number of 12 subjects for pilot studies.

To avoid confounding by BMI and age, patients will be matched for BMI and age to ensure an equal distribution between the groups of the variables believed to be confounding. Patients will not be blinded to study condition assignment.

ELIGIBILITY:
Inclusion Criteria:

* both sexes
* age 18-65 yrs
* BMI > 35 kg/m2

Exclusion Criteria:

* severe psychiatric conditions
* acute respiratory disease
* acute cardiovascular disease
* unstable hypertension
* cold intolerance
* claustrophobia
* pregnancy
* recent modification of usual drug treatment
* previous treatment with WBC
* weight loss in the last 3 months
* body temperature greater than 37.5°C.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline blood catecholamine levels (epinephrine, norepinephrine and dopamine) | up to 3 weeks
  Catecholamine levels (ng/ml) in plasma samples will be measured at baseline and two weeks later, after multidisciplinary rehabilitation (R group) or multidisciplinary rehabilitation + WBC (RWBC group).

SECONDARY OUTCOMES:
Change in skin temperatures after every session of WBC | up to 1 minute
  The change in skin temperature of all body regions considered will be measured (nape of the neck, right quadriceps, right popliteal fossa, right calf) within 1 minute before and 1 minute after every session of WBC.
Change from baseline biochemical blood parameters HDL, LDL, Triglycerides and Glucose | up to 4 weeks
  Analysis of blood biochemical parameters HDL, LDL, Triglycerides and Glucose (mg/dl) at baseline and two weeks later, after multidisciplinary rehabilitation (R group) or multidisciplinary rehabilitation + WBC (RWBC group).
Change from baseline biochemical blood parameter HBA1C% | up to 4 weeks
  Analysis of HBA1C% at baseline and two weeks later, after multidisciplinary rehabilitation (R group) or multidisciplinary rehabilitation + WBC (RWBC group).
Change from baseline systolic blood pressure and diastolic blood pressure (mmHg) | up to 4 weeks
  Measurement of systolic blood pressure (PAS), diastolic blood pressure (PAD) at baseline and two weeks later, after multidisciplinary rehabilitation (R group) or multidisciplinary rehabilitation + WBC (RWBC group).
Change from baseline heart rate variability (HRV) (bpm) | up to 4 weeks
  Measurement of hear rate (HR) at baseline and two weeks later, after multidisciplinary rehabilitation (R group) or multidisciplinary rehabilitation + WBC (RWBC group).
Change from baseline weight | up to 4 weeks
  Measurement of Weight (kg) at baseline and two weeks later, after multidisciplinary rehabilitation (R group) or multidisciplinary rehabilitation + WBC (RWBC group).
Change from baseline BMI | up to 4 weeks
  Measurement of BMI (kg/m2) at baseline and two weeks later, after multidisciplinary rehabilitation (R group) or multidisciplinary rehabilitation + WBC (RWBC group).
Change from baseline waist circumference | up to 4 weeks
  Measurement of waist circumference (cm) at baseline and two weeks later, after multidisciplinary rehabilitation (R group) or multidisciplinary rehabilitation + WBC (RWBC group).
Change from baseline % of Fat Mass (FM), Free Fat Mass (FFM) and Muscle Mass (MM) | up to 4 weeks
  Measurement of FM, MM and FFM % at baseline and two weeks later, after multidisciplinary rehabilitation (R group) or multidisciplinary rehabilitation + WBC (RWBC group).
Change from baseline aerobic endurance | up to 4 weeks
  Measurement of aerobic endurance using the six-minute walk test (m) at baseline and two weeks later, after multidisciplinary rehabilitation (R group) or multidisciplinary rehabilitation + WBC (RWBC group).
Change from baseline balance and functional mobility | up to 4 weeks
  Measurement of balance and functional mobility using the Timed Up and Go test (sec) at baseline and two weeks later, after multidisciplinary rehabilitation (R group) or multidisciplinary rehabilitation + WBC (RWBC group).
Change from baseline isometric strength | up to 4 weeks
  Measurement of isometric strength using the hand grip test (kg) at baseline and two weeks later, after multidisciplinary rehabilitation (R group) or multidisciplinary rehabilitation + WBC (RWBC group).
Change from baseline of subjective well-being | up to 12 months
  Patients' subjective well-being was assessed using the World Health Organization's self-administered questionnaire: Five Well-Being Index (WHO-5). The raw score ranges from 0 to 25, where 0 represents the worst possible quality of life and 25 represents the best possible quality of life.
Change from baseline of subjective psychological well-being | up to 12 months
  Patients' subjective psychological well-being was assessed using the Psychological General Well-Being Index (PGWBI), a 22-item self-report questionnaire designed to measure subjective well-being or distress over the past 28 days. The items reflect the six subscales: anxiety, depression, positive well-being, self-control, general health and vitality, comprising 5, 3, 4, 3, 3 and 4 items, respectively. A 6-point Likert scale (0 to 5) provides a total and subscale score of up to 110 points, where higher scores indicate better PGWB. PGWBI scores were grouped into the following categories: 0-60 Severe Distress, 61-71 Moderate Distress, 72-92 No Distress, and 93-110 PWB.
Change from baseline of the obesity-related disability | up to 12 months
  Obesity-related disability is assessed using the Test of Obesity-Related Disability (SIO Obesity-Related Disability Test, TSD-OC). The TSD-OC consists of 7 sections with a total of 36 items exploring the following dimensions of disability: pain, stiffness, ADL and mobility in the home, activities in the home, activities outside the home, work activities, and social life.
  The patient is asked to subjectively rate the disability for each item by means of a visual analog scale (VAS): a value of 10 indicates the highest level of disability and a value of 0 the absence of difficulty in performing that particular function. A person's degree of disability is assessed by relating the score obtained to the maximum score obtainable (360). A person is considered disabled if he or she has a disability score greater than 33% or has a score ≥8/10 in any of the items.
Change from baseline of the impact of fibromyalgia | up to 12 months
  The FIQ is scored in such a way that a higher score indicates a greater impact of the syndrome on the person. Each of the 10 items has a maximum possible score of 10. Thus, the maximum possible score is 100. The average score for a patient with fibromyalgia is about 50; patients with severe conditions usually have a score of more than 70.
Change from baseline of the conditions of patients with hip and knee osteoarthritis | up to 12 months
  Patients are asked to fill out the Western Ontario and McMaster Universities Osteoarthritis index (WOMAC, only for patients with osteoarthritis). The score obtained varies from 0 to 96 depending on the symptomatology described. Statistical analysis of the WOMAC values before and after the considered treatments allows us to evaluate the effectiveness of the treatments.
Change from baseline of subjective sleep quality | up to 12 months
  Patients' subjective improvement in sleep quality is assessed using the following self-administered questionnaires: Pittsburgh sleep quality index (PSQI).
  In scoring the PSQI, seven component scores are derived, each scored 0 (no difficulty) to 3 (severe difficulty). The component scores are summed to produce a global score (range 0 to 21). Higher scores indicate worse sleep quality.
Change from baseline of subjective pain level | up to 12 months
  Subjective pain level improvement is measured using the Pain Numeric Rating Scale (PNRS). The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable").
Change from baseline of chronic pain | up to 12 months
  Chronic pain improvement is measured only in patients with chronic pain using the Brief Pain Inventory (BPI). The BPI measures how much pain has interfered with seven daily activities, including general activity, walking, work, mood, enjoyment of life, relations with others, and sleep. BPI pain interference is typically scored as the mean of the seven interference items.
  The BPI scale defines pain as follows: Worst Pain Score: 1 - 4 = Mild Pain. Worst Pain Score: 5 - 6 = Moderate Pain. Worst Pain Score: 7 - 10 = Severe Pain.
Change from baseline of the use of pain medications | up to 12 months
  The use of pain medications is assessed using the Quantitative Analgesic Questionnaire (QAQ) is a instrument designed to comprehensively document patient-reported medication use, generate scores to quantify it (by individual drug, class, and/or overall), and compare it (qualitatively and/or quantitatively) to the regimen as prescribed.
Change from baseline of subjective fatigue perception | up to 12 months
  The impact of fatigue on patients was evaluated using the fatigue severity scale (FSS). The raw score ranges from 9 to 63. A total score of less than 36 suggests that the subject may not be suffering from fatigue while a total score of 36 or more suggests further evaluation by a physician.
  Based on the frequency of episodes, a score of 0 to 4 points is given for the reported parameters up to a maximum of 20 (severe fecal incontinence) to obtain which all steps considered must be indicated and summed
Change from baseline of the subjective quantification of the fear of movement | up to 12 months
  The quantification of the fear of movement is assessed using the Tampa Scale of Kinesiophobia (TSK-I).
  The TSK is a self-completed questionnaire and the range of scores are from 17 to 68 where the higher scores indicate an increasing degree of kinesiophobia.
Change from baseline in depression | up to 12 months
  Depression is assessed using the Beck Depression Inventory (BDI). The highest positive score can be 63, the lowest 0. The standard cut-off scores were as follows: 0-9: indicates minimal depression. 10-18: indicates mild depression. 19-29: indicates moderate depression.
  The highest positive score can be 63, the lowest 0. The cut-off is 17 points.
Change from baseline in anxiety | up to 12 months
  Anxiety is assessed using the State-Trait Anxiety Inventory (STAI). Scores range from 20 to 80, with higher scores correlating with greater anxiety.
Change from baseline in the sleep condition | up to 12 months
  Sleep condition is assessed using the Sleep Condition Indicator (SCI). Scores range from 0 to 32 with scores ≤ 16 considered indicative of insomnia disorder in the general population Sleep condition is assessed using the Sleep Condition Indicator (SCI). Scores range from 0 to 32.
Change from baseline of subjective sleepiness | up to 12 months
  Patients' subjective sleepiness is assessed using the Epworth Sleepiness Scale. The test is a list of eight situations in which you rate your tendency to become sleepy on a scale of 0, no chance of dozing, to 3, high chance of dozing. 1 to 6 points: Normal sleep; 7 to 8 points: Average sleepiness; 9 to 24 points: Abnormal (possibly pathologic) sleepiness.
Change from baseline in Depression, Anxiety and Stress | up to 12 months
  Depression, anxiety and stress are assessed using the Depression, Anxiety and Stress Scale - 21 Items (DASS-21). Scores range from 0 to 32 for every item (Depression, Anxiety and Stress). The total score represents overall distress (0 to 30), with higher scores indicating more severe distress or a greater number of symptoms. Two subscales are presented: Anxiety-Stress: Items 1, 4, 6, 7, 8, 9 (raw score range = 0 to 18) Depression: Items 2, 3, 5, 10 (raw score range = 0 to 12)
Change from baseline in Central Sensitization Inventory (CSI) | up to 12 months
  Central Sensitization Inventory is a self-report outcome measure designed to identify patients who have symptoms that may be related to Central Sensitisation (CS) or central sensitivity syndromes (CSS). Responses are recorded about the frequency of each symptom, with a Likert scale from 0 (never) to 4 (always), resulting in a total possible score of 100. Higher scores are associated with a higher degree of self-reported symptomology.
Change from baseline in intestinal function | up to 12 months
  Constipation symptoms are assessed using the Wexner score. Based on the frequency of episodes, a score of 0 to 4 points is given for the reported parameters up to a maximum of 20 (severe fecal incontinence) to obtain which all steps considered must be indicated and summed
Follow-up questionnaires or telephone interviews | up to 12 months
  The subjective improvement of patients is assessed through the administration of questionnaires or follow-up telephone interviews on general health and well-being, quality of life, sleep quality, pain level, use of medications, fatigue and psychological aspects (i.e. depression and anxiety).
Change from baseline Sleep Disturbance | up to 12 months
  Patients' sleep disturbance is assessed using the PROMIS Sleep Disturbance Short Form survey. Each item on the measure is rated on a 5-point scale (1=never; 2=rarely; 3=sometimes; 4=often; and 5=always) with a range in score from 8 to 40 with higher scores indicating greater severity of sleep disturbance.
Change from baseline Global Health | up to 12 months
  Patients' global health is assessed using the PROMIS Global Health Scale. The possible score ranges from 0 to 20 points in each case. 0 points represent the patient's most severe physical and/or mental impairment, while 20 points represent the best possible state of health.
Change from baseline health status | up to 12 months
  Patients are asked to fill out Short Form 36, a questionnaire constructed to detect health status. Each item on the questionnaire is rated, and a higher number indicates that the person enjoys better overall health. In addition, each item is rated on a scale of 0 to 100, with 0 and 100 being the lowest and highest possible scores. The scores indicate the percentage of the possible score that was actually achieved.

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Capodaglio, Prof, MD, Principal Investigator — IRCCS Istituto Auxologico Italiano
Locations (1):
- IRCCS Istituto Auxologico Italiano Ospedale San Giuseppe, Oggebbio, Verbano-Cusio-Ossola, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thorp AA, Schlaich MP. Relevance of Sympathetic Nervous System Activation in Obesity and Metabolic Syndrome. J Diabetes Res. 2015;2015:341583. doi: 10.1155/2015/341583. Epub 2015 Apr 30. PMID 26064978
- [Background] Qi Z, Ding S. Obesity-associated sympathetic overactivity in children and adolescents: the role of catecholamine resistance in lipid metabolism. J Pediatr Endocrinol Metab. 2016 Feb;29(2):113-25. doi: 10.1515/jpem-2015-0182. PMID 26488603
- [Background] Fisher JP, Young CN, Fadel PJ. Central sympathetic overactivity: maladies and mechanisms. Auton Neurosci. 2009 Jun 15;148(1-2):5-15. doi: 10.1016/j.autneu.2009.02.003. Epub 2009 Mar 6. PMID 19268634
- [Background] Grassi G, Biffi A, Seravalle G, Trevano FQ, Dell'Oro R, Corrao G, Mancia G. Sympathetic Neural Overdrive in the Obese and Overweight State. Hypertension. 2019 Aug;74(2):349-358. doi: 10.1161/HYPERTENSIONAHA.119.12885. Epub 2019 Jun 17. PMID 31203727
- [Background] Fontana JM, Bozgeyik S, Gobbi M, Pitera P, Giusti EM, Dugue B, Lombardi G, Capodaglio P. Whole-body cryostimulation in obesity. A scoping review. J Therm Biol. 2022 May;106:103250. doi: 10.1016/j.jtherbio.2022.103250. Epub 2022 May 4. PMID 35636880
- [Background] White GE, Wells GD. Cold-water immersion and other forms of cryotherapy: physiological changes potentially affecting recovery from high-intensity exercise. Extrem Physiol Med. 2013 Sep 1;2(1):26. doi: 10.1186/2046-7648-2-26. PMID 24004719
- [Background] Hanssen MJ, van der Lans AA, Brans B, Hoeks J, Jardon KM, Schaart G, Mottaghy FM, Schrauwen P, van Marken Lichtenbelt WD. Short-term Cold Acclimation Recruits Brown Adipose Tissue in Obese Humans. Diabetes. 2016 May;65(5):1179-89. doi: 10.2337/db15-1372. Epub 2015 Dec 30. PMID 26718499
- [Background] Wiecek M, Szymura J, Sproull J, Szygula Z. Whole-Body Cryotherapy Is an Effective Method of Reducing Abdominal Obesity in Menopausal Women with Metabolic Syndrome. J Clin Med. 2020 Aug 30;9(9):2797. doi: 10.3390/jcm9092797. PMID 32872598
- [Background] Lombardi G, Ziemann E, Banfi G. Whole-Body Cryotherapy in Athletes: From Therapy to Stimulation. An Updated Review of the Literature. Front Physiol. 2017 May 2;8:258. doi: 10.3389/fphys.2017.00258. eCollection 2017. PMID 28512432
- [Background] Costello JT, Baker PR, Minett GM, Bieuzen F, Stewart IB, Bleakley C. Whole-body cryotherapy (extreme cold air exposure) for preventing and treating muscle soreness after exercise in adults. Cochrane Database Syst Rev. 2015 Sep 18;2015(9):CD010789. doi: 10.1002/14651858.CD010789.pub2. PMID 26383887
- [Background] Smolander J, Westerlund T, Uusitalo A, Dugue B, Oksa J, Mikkelsson M. Lung function after acute and repeated exposures to extremely cold air (-110 degrees C) during whole-body cryotherapy. Clin Physiol Funct Imaging. 2006 Jul;26(4):232-4. doi: 10.1111/j.1475-097X.2006.00675.x. PMID 16836696
- [Background] Banfi G, Melegati G, Barassi A, d'Eril GM. Effects of the whole-body cryotherapy on NTproBNP, hsCRP and troponin I in athletes. J Sci Med Sport. 2009 Nov;12(6):609-10. doi: 10.1016/j.jsams.2008.06.004. Epub 2008 Oct 2. PMID 18835219
- [Background] Gobbi M, Trotti G, Tanzi M, Kasap F, Pitera P, Capodaglio P. POST-COVID SYMPTOMS AND WHOLE-BODY CRYOTHERAPHY: A CASE REPORT. J Rehabil Med Clin Commun. 2022 Jan 13;5:1000075. doi: 10.2340/20030711-1000075. eCollection 2022. No abstract available. PMID 35154582
- [Background] Varallo G, Pitera P, Fontana JM, Gobbi M, Arreghini M, Giusti EM, Franceschini C, Plazzi G, Castelnuovo G, Capodaglio P. Is Whole-Body Cryostimulation an Effective Add-On Treatment in Individuals with Fibromyalgia and Obesity? A Randomized Controlled Clinical Trial. J Clin Med. 2022 Jul 26;11(15):4324. doi: 10.3390/jcm11154324. PMID 35893415
- [Background] Alito A, Fontana JM, Franzini Tibaldeo E, Verme F, Pitera P, Miller E, Cremascoli R, Brioschi A, Capodaglio P. Whole-Body Cryostimulation in Multiple Sclerosis: A Scoping Review. J Clin Med. 2024 Mar 29;13(7):2003. doi: 10.3390/jcm13072003. PMID 38610768
- [Derived] Cerfoglio S, Verme F, Fontana JM, Alito A, Galli M, Capodaglio P, Cimolin V. Effects of whole-body cryostimulation on spinal and shoulder range of motion in individuals with obesity. Front Rehabil Sci. 2025 Jul 23;6:1568280. doi: 10.3389/fresc.2025.1568280. eCollection 2025. PMID 40772266